CLINICAL TRIAL: NCT06923592
Title: Serological Testing and Treatment for Plasmodium Vivax Malaria: a Cluster-Randomised Trial in Ethiopia and Madagascar
Brief Title: Serological Testing and Treatment for Plasmodium Vivax Malaria: a Trial in Ethiopia and Madagascar
Acronym: PvSTATEM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Institut Pasteur (Industry); Institut Pasteur de Madagascar (Other); Armauer Hansen Research Institute (AHRI), Ethiopia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 29643
Record Dates: First submitted 2025-04-03; First posted 2025-04-11 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-06

CONDITIONS: Malaria Vivax; Malaria Falciparum; Plasmodium Vivax; Plasmodium Falciparum
Keywords: Plasmodium vivax; Vivax; PvSeroTAT; PvSTATEM; Primaquine; serology; Cluster randomised trial; G6PD
MeSH Terms: conditions — Malaria, Vivax; Malaria, Falciparum

STUDY DESIGN:
Intervention Model Description: In each country, 24 clusters (48 clusters in total) will be randomly allocated to one of the two interventions: Arm 1 (PvSeroTAT intervention) or Arm 2 (Control arm). Within each cluster, approximately 400 participants (range 100-600) that fulfill the inclusion and exclusion criteria will be enrolled. At baseline (month 0) and month 6 serology for P. vivax infections will be performed in all study participants. In the clusters in the PvSeroTAT arm, participants with a positive P. vivax serology at baseline or month 6 will be treated with 7 days of primaquine 0.5mg/kg/day and a three-day course of either chloroquine (Ethiopia) or artesunate-amodiaquine (Madagascar).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PvSeroTAT intervention (Experimental)
  Interventions: Combination Product: PvSeroTAT
- Control arm (Other)
  Interventions: Diagnostic Test: Control

INTERVENTIONS:
Combination Product: PvSeroTAT — Two rounds (month 0 and month 6) of serological screening for antibodies against P. vivax in the blood of all eligible cluster inhabitants. In the clusters in the PvSeroTAT arm, participants with a positive P. vivax serology at baseline or month 6 will be treated with 7 days of primaquine 0.5mg/kg/day and a three-day course of either chloroquine (Ethiopia) or artesunate-amodiaquine (Madagascar).
  Arms: PvSeroTAT intervention
Diagnostic Test: Control — Two rounds (month 0 and month 6) of serological screening for antibodies against P. vivax in the blood of a subset of eligible cluster inhabitants. Serological status will be assessed at a later stage (months later) and will not lead to treatment of sero-positive individuals.
  Arms: Control arm

SUMMARY:
The resilience of P. vivax to malaria elimination efforts is due to its ability to form dormant liver stages (hypnozoites) that reactivate weeks to months after the initial infection causing recurrent episodes of malaria (relapses) and ongoing parasite transmission. Relapses account for a majority of recurrent infections and clinical cases of P. vivax malaria, and therefore have a significant effect on morbidity at the individual level.

With current technology, it is not possible to directly measure hypnozoite biomarkers. Rather than directly detecting hypnozoites, our team developed an indirect approach by measuring antibodies induced by the primary blood-stage infection. Antibodies to different blood-stage antigens decay at different rates. Measuring antibodies to a carefully selected panel of P. vivax antigens can aid to identify individuals who have been infected within the previous 9 months (approximately the lifespan of hypnozoites).

A serological test based on selected P. vivax antigens can detect recent exposure and predict future relapses. Coupling this test with a safe and efficacious primaquine treatment regimen, results in a population-based intervention to target the hypnozoite reservoir. This intervention is referred to as Plasmodium vivax Serological Testing and Treatment (PvSeroTAT).

PvSTATEM is a cluster randomised trial in Madagascar and Ethiopia. This study will provide insights into the feasibility, acceptability, and efficacy of the PvSeroTAT approach. In this study, individuals, randomised by clusters, will be tested for the presence of serological markers of a recent P. vivax infection, followed by a targeted drug treatment intervention aimed at killing P. vivax hypnozoites.

DETAILED DESCRIPTION:
In each country, 24 clusters (48 clusters in total) will be randomly allocated using computer generated numbers to one of the two interventions:

Arm 1 (PvSeroTAT intervention) or Arm 2 (Control arm). Within each cluster, approximately 400 participants (range 100-600) will be enrolled, based on the trial's inclusion and exclusion criteria. At baseline (month 0) and month 6 serology for P. vivax infections will be performed in all study participants. In the clusters in the PvSeroTAT arm, participants with a positive P. vivax serology at baseline or month 6 will be approached for treatment. First G6PD enzyme activity will be measured. If the enzyme activity is normal and no other contra-indication for treatment are found, the participants will be treated with 7 days of primaquine 0.5mg/kg/day and a three-day course of either chloroquine (Ethiopia) or artesunate-amodiaquine (Madagascar). It is possible that a participant could receive a radical P. vivax treatment at both baseline (month 0) and month 6. Participants will be monitored for side effects and adherence during the first 7 days after the start of antimalarial treatments. In addition, blood samples will be taken to measure hemoglobin levels to monitor for post-treatment hemolysis.

In the clusters in both arms, the incidence of malaria will be monitored through passive case detection in health posts up to 18 months after the first intervention. All cases that are detected during the passive case detection will be treated according to the national guidelines.

At month 12 and month 18 of the study, a cross sectional survey will be conducted in all study clusters. Blood samples will be taken to determine the prevalence of P. vivax and P. falciparum through PCR assays.

ELIGIBILITY:
Inclusion Criteria:

* Participant will remain in the study area for at least the next month.
* Participant is older than 12 months

Exclusion Criteria:

• Participant is unwilling to participate.

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19200 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2027-04-28 (Estimated); Study Completion 2027-04-28 (Estimated)

PRIMARY OUTCOMES:
Proportion of individuals with PCR detectable P. vivax blood-stage infections 6 months after the second round of PvSeroTAT or 6 months after the second round of blood sampling in the control clusters. | 6 months after the second round of PvSeroTAT or 6 months after the second round of blood sampling in the control clusters.
  6 months after the second round of PvSeroTAT, a blood sample will be collected from participants through fingerprick in the intervention clusters. In the control clusters a blood sample to determine PCR prevalence will be collected 6 months after the second round of blood sampling in that control cluster.

SECONDARY OUTCOMES:
Proportion of individuals with PCR detectable P. vivax blood-stage infections 12 months after the second round of PvSeroTAT or 12 months after the second round of blood sampling in the control clusters. | 12 months after the second round of PvSeroTAT or 12 months after the second round of blood sampling in the control clusters.
  12 months after the second round of PvSeroTAT, a blood sample will be collected from participants through fingerprick in the intervention clusters. In the control clusters a blood sample to determine PCR prevalence will be collected 12 months after the second round of blood sampling in that control cluster.
Proportion of individuals with PCR detectable P. vivax blood-stage infections 6 months after the first round of PvSeroTAT (before second round) or 6 months after the first round of blood sampling in the control clusters. | 6 months after the first round of PvSeroTAT or 6 months after the first round of blood sampling in the control clusters.
  6 months after the first round of PvSeroTAT, a blood sample will be collected from participants through fingerprick in the intervention clusters. In the control clusters a blood sample to determine PCR prevalence will be collected 6 months after the first round of blood sampling in that control cluster.
Decrease of mean cluster prevalence of PCR detectable P. vivax blood-stage infections at month 6 after the first round of PvSeroTAT or 6 months after the first round of blood sampling in the control clusters, compared to baseline. | 6 months after the first round of PvSeroTAT or 6 months after the first round of blood sampling in the control clusters.
Decrease of mean cluster prevalence of PCR detectable P. vivax blood-stage infections at month 12 after the first round of PvSeroTAT or 12 months after the first round of blood sampling in the control clusters, compared to baseline. | 12 months after the first round of PvSeroTAT or 12 months after the first round of blood sampling in the control clusters.
Decrease of mean cluster prevalence of PCR detectable P. vivax blood-stage infections at month 18 after the first round of PvSeroTAT or 18 months after the first round of blood sampling in the control clusters, compared to baseline. | 18 months after the first round of PvSeroTAT or 18 months after the first round of blood sampling in the control clusters.
Incidence of clinical cases of P. vivax and P. falciparum malaria during the 6 months after the first round of PvSeroTAT or during the 6 months after the first round of blood sampling in the control clusters. | 6 months after the first round of PvSeroTAT or 6 months after the first round of blood sampling in the control clusters.
Incidence of clinical cases of P. vivax and P. falciparum malaria during the 12 months after the first round of PvSeroTAT or during the 12 months after the first round of blood sampling in the control clusters. | 12 months after the first round of PvSeroTAT or 12 months after the first round of blood sampling in the control clusters.
Incidence of clinical cases of P. vivax and P. falciparum malaria during the 18 months after the first round of PvSeroTAT or during the 18 months after the first round of blood sampling in the control clusters. | 18 months after the first round of PvSeroTAT or 18 months after the first round of blood sampling in the control clusters.
Hemoglobin level at day 3 | Day 3
Hemoglobin level at day 7 | Day 7
Decrease in Hemoglobin between baseline and day 3 (absolute and proportional) | Day 3
Decrease in Hemoglobin between baseline and day 7 (absolute and proportional) | Day 7
Incidence of potential signs of clinically relevant Haemolysis | 7 days
  25% drop in hemoglobin or hemoglobin<7gram/dL or macroscopic haemoglobinuria or the need for a blood transfusion
Incidence of Serious Adverse Events | 18 months after the first round of PvSeroTAT or 18 months after the first round of blood sampling in the control clusters.
Coverage of serological tests for P. vivax antibodies as proportion of number of individuals per cluster | Day 0 of month 0 or month 6
Proportion of eligible individuals that refuses participation in the study | Day 0 of month 0 or month 6
Proportion of participants with positive P. vivax serology that refuses P. vivax treatment | Day 1 of drug administration
Proportion of serological positive individuals that start primaquine treatment | Day 1 of drug administration
Proportion of study participants that complete the 7-day course of primaquine treatment. | Day of start of treatment until day 7 of treatment
Proportion of individuals that vomits at least once within 1 hour after treatment | Day of start of treatment until day 7 of treatment
Proportion of individuals that vomits twice within 1 hour after treatment. | Day of start of treatment until day 7 of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Chris Drakeley, Principal Investigator — London School of Hygiene and Tropical Medicine; Michael T White, Principal Investigator — Institut Pasteur; Rindra Randremanana, Principal Investigator — Institut Pasteur de Madagascar; Fitsum G Tadesse, Principal Investigator — Armauer Hansen Research Institute
Locations (2):
- Armauer Hansen Research Institute, Addis Ababa, Ethiopia
- Institut Pasteur de Madagascar, Antananarivo, Madagascar

IPD SHARING:
Plan to Share IPD: Yes
Anonymised demographic data (e.g. age and sex). P. vivax serology results. Clinical parameters such as hemoglobin levels and clinical symptoms. Results of PCR assays for Plasmodium vivax and Plasmodium falciparum.
Supporting Information: Study Protocol, SAP
Time Frame: After publication of the manuscripts detailing the results of the study.

REFERENCES:
- See also: PvSTATEM project website — https://www.pvstatem.eu